CLINICAL TRIAL: NCT02977026
Title: Comparing the Efficacy of the Alcohol Help Centre and Check Your Drinking to a no Intervention Control Condition: Randomized Controlled Trial
Brief Title: Comparing the Efficacy of the Alcohol Help Centre and Check Your Drinking to a no Intervention Control Condition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, John Cunningham, Senior Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 107/2016
Record Dates: First submitted 2016-11-27; First posted 2016-11-30 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Alcohol Consumption
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (No Intervention): A questionnaire that asks individuals what components of an online intervention they might find useful.
- Check Your Drinking (CYD) (Experimental): Internet based program of lower intensity as compared to the "Alcohol Help Centre. It was designed to provide personalized normative feedback aimed at motivating reductions in drinking
  Interventions: Behavioral: CYD
- Alcohol Help Centre (AHC) (Experimental): Internet based program of higher intensity as compared to the "Check Your Drinking" intervention. It was designed to assesses drinking patterns, increase self-awareness of individual triggers, and set and achieve goals regarding drinking.
  Interventions: Behavioral: AHC

INTERVENTIONS:
Behavioral: CYD
  Arms: Check Your Drinking (CYD)
Behavioral: AHC
  Arms: Alcohol Help Centre (AHC)

SUMMARY:
Alcohol is one of the leading contributors to premature mortality and disability. Most people with alcohol problems will never seek treatment. There is a need to develop alternate ways to help problem drinkers outside of formal treatment settings.

One promising strategy is Internet-based interventions for problem drinkers. Our recently completed RCT comparing a brief (Check Your Drinking; CYD) versus an extended (Alcohol Help Centre; AHC) Internet intervention for problem drinkers found that, while there was a reduction in drinking across time for both interventions, there was no significant (p > .05) difference in reductions in drinking between the two interventions. Based on these results, it is not justifiable to say that either intervention 'worked' as there was no comparison condition of participants who received no active intervention. The current trial proposes to address this limitation by conducting an RCT comparing the CYD, AHC, and a no intervention control condition.

Participants will be recruited through Amazon's MTurk crowdsourcing platform. Participants identified as problem drinkers based on an initial survey will be invited to complete another survey in 6 months time. Those who are interested will be randomized to receive access to the Check Your Drinking screener (CYD condition), Alcohol Help Centre (AHC condition) or a feedback questionnaire (control condition). At six-months post-baseline, the MTurk portal will be used to send invitation emails that contain a link to the follow-up survey. The primary hypothesis to be tested is that participants receiving access to the AHC intervention will report a greater reduction in AUDIT-C scores and in number of drinks in a typical week than participants in the CYD intervention. Further, participants in the CYD condition will report a greater level of reduction AUDIT-C scores and in number of drinks in a typical week between the baseline survey and six-month follow-up as compared to participants in the no intervention control condition.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or over
* A score of 8 or over on the Alcohol Use Disorders Identification Test (AUDIT)
* Typically consumes 15 or more drinks per week,
* Willingness to complete a 6-month follow-up survey

Exclusion Criteria:None

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2016-12; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change in number of drinks in a typical week from baseline | 6 months
  Sum of number of drinks consumed in a typical week

CONTACTS AND LOCATIONS:
Overall Officials: John A Cunningham, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Godinho A, Schell C, Cunningham JA. How one small text change in a study document can impact recruitment rates and follow-up completions. Internet Interv. 2019 Oct 20;18:100284. doi: 10.1016/j.invent.2019.100284. eCollection 2019 Dec. PMID 31890631
- [Derived] Cunningham JA, Godinho A, Bertholet N. Outcomes of two randomized controlled trials, employing participants recruited through Mechanical Turk, of Internet interventions targeting unhealthy alcohol use. BMC Med Res Methodol. 2019 Jun 14;19(1):124. doi: 10.1186/s12874-019-0770-4. PMID 31200648